CLINICAL TRIAL: NCT05922761
Title: An Open-Label, Phase 2 Study to Evaluate the Activity of Belumosudil in Subjects With New Onset and Incipient Bronchiolitis Obliterans Syndrome Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: BElumosudil for Bronchiolitis Obliterans Prevention/Therapy (BEBOP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Sanofi (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Corey S. Cutler, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-043
Record Dates: First submitted 2023-06-03; First posted 2023-06-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans; Lung Diseases; Chronic Graft Versus Host Disease
Keywords: Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans; Lung Disease; Allogeneic hematopoietic stem cell transplant; HSCT; Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Bronchiolitis Obliterans; Lung Diseases | interventions — belumosudil; KD025; acetamide; Fluticasone; Azithromycin; Prednisone; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: Belumosudil + Standard of Care Medications (Experimental): 30 participants with bronchiolitis obliterans syndrome (BOS) will complete study procedures as follows:
  * Drug diary
  * CT scans at Cycles 3 and 7 and at End of Treatment.
  * Cycle 1
    * Day 1 - 28 of 28-day cycle: Predetermined dose of Belumosudil 1x daily.
    * Predetermined doses of Fluticasone, Montelukast, and Prednisone 1x daily.
    * Predetermined dose of azithromycin 3 days per treatment week.
  * Cycle 2 - 3
    * Day 1 - 28 of 28-day cycle: Predetermined dose of Belumosudil 1x daily.
    * Predetermined doses of Fluticasone Montelukast 1x daily. Predetermined doses of Prednisone 1x daily at treating physician's discretion.
    * Predetermined dose of azithromycin 3 days per treatment week.
  * Cycle 4 - 12
    * Day 1 - 28 of 28-day cycle: Predetermined dose of Belumosudil 1x daily.
    * Predetermined doses of Fluticasone and Montelukast 1x daily.
    * Predetermined dose of azithromycin 3 days per treatment week.
  Interventions: Drug: Belumosudil; Drug: Fluticasone; Drug: Azithromycin; Drug: Prednisone; Drug: Montelukast
- Cohort B: Belumosudil (Experimental): 15 participants with signs concerning developing BOS will complete study procedure as follows:
  * Drug diary
  * CT scans at Cycles 3 and 7 and at End of Treatment.
  * Cycle 1 - 12 - Day 1 - 28 of 28-day cycle: Predetermined dose of Belumosudil 1x daily.
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Kinase inhibitor, tablet taken orally
  Other Names: Rezurock, KD025, 2-{3-[4-(1H-indazol-5-ylamino)-2-quinazolinyl]phenoxy}-N-(propan-2-yl) acetamide, C26H24N6O2
Drug: Fluticasone — Via inhalation by metered-dose inhaler.
  Other Names: Fluticasone Propionate
  Arms: Cohort A: Belumosudil + Standard of Care Medications
Drug: Azithromycin — Semi-synthetic macrolide antibiotic, taken orally
  Other Names: Zithromax
  Arms: Cohort A: Belumosudil + Standard of Care Medications
Drug: Prednisone — Corticosteroid, taken orally
  Arms: Cohort A: Belumosudil + Standard of Care Medications
Drug: Montelukast — Leukotriene Receptor Antagonist, taken orally
  Other Names: Singulair
  Arms: Cohort A: Belumosudil + Standard of Care Medications

SUMMARY:
The goal of this research study is to test the efficacy of a novel immunosuppressive agent, belumosudil, in allogeneic hematopoietic stem cell transplant (HSCT) recipients who have been newly diagnosed or have developing (early stage) bronchiolitis obliterans syndrome (BOS).

The name of the study drugs involved in this study are:

* Belumosudil (an immunotherapy)
* Fluticasone (an intranasal corticosteroid)
* Azithromycin (an antibiotic)
* Montelukast (a leukotriene receptor antagonist)
* Prednisone (a corticosteroid)

DETAILED DESCRIPTION:
This is an open-label, single-arm, single-stage phase 2 study to evaluate the activity of Belumosudil in subjects with new onset of bronchiolitis obliterans syndrome (BOS) (Cohort A) and for subjects with incipient BOS (Cohort B) following allogeneic hematopoietic cell transplantation (HCT). Belumosudil is a novel immunosuppressive agent that has both immunosuppressive activity as well as antifibrotic (slowing down the rate of fibrosis or scarring in the lungs) properties.

Participants will be placed into one of two treatment groups: Group A Belumosudil + standard of care medications for BOS versus Group B Belumosudil only.

The U.S. Food and Drug Administration (FDA) has not approved belumosudil for the initial or preventative therapy of BOS, but it has been approved for the treatment of Chronic Graft Versus Host Disease (cGVHD).

The other study drugs, Fluticasone, Azithromycin, Montelukast, and Prednisone are FDA approved as standard of care drugs for BOS.

Study procedures include screening for eligibility, treatment visits, blood tests, pulmonary function tests, bronchoscopy wit bronchoalveolar lavage, and Computed Tomography (CT) Scans.

Participants will receive study treatment for 11 months (48 weeks) and will be followed for an additional 12 months after completion of study treatment.

It is expected that about 45 people (30 in Group A and 15 in Group B) will take part in this research study.

The National Heart, Lung, and Blood Institute (NHLBI) is supporting this research study by providing funding.

Sanofi is supporting this research study by providing study drug, Belumosudil.

ELIGIBILITY:
Inclusion Criteria Cohort A:

* Diagnosis of BOS after HCT using pulmonary function testing, per the NIH diagnostic criteria17 OR the Atypical BOS criteria33 3.1.2.1 NIH Diagnostic Criteria for BOS. All of the following must be met:

  * FEV1/VC < 0.7 or <5th percentile of predicted (FEV1 = Forced Expiratory Volume in 1 second; VC = Vital Capacity (either FVC, Forced Vital Capacity, or SVC, Slow Vital Capacity, whichever is greater)
  * FEV1 <75% of predicted with ≥ 10% absolute decline over less than 2 years. FEV1 should not correct to >75% of predicted with albuterol, and the absolute decline for the corrected values should still remain ≥ 10% over 2 years.
  * Absence of active infection in the respiratory tract, documented with investigations directed by clinical symptoms, such as chest radiographs or computed tomographic scans or microbiologic cultures (sinus aspiration, upper respiratory tract viral screen, sputum culture, bronchoalveolar lavage).
  * One of the two supporting features of BOS:

    * i - Evidence of air trapping by expiratory CT or small airway thickening or bronchiectasis by high-resolution chest CT OR
    * ii - Evidence of air trapping by PFTs: RV (Residual Volume) > 120% of predicted or RV/TLC elevated outside the 90% confidence interval (RV/Total Lung Capacity).
* Atypical Criteria for BOS:

  * FEV1 <80% of predicted with ≥ 10% absolute decline over the last 2 years or since transplant. The remote comparator can be an evaluation of PFTs done within 2 years of the PFTs assessment being evaluated to determine eligibility or the PFT assessment done prior to transplant.
  * VC < 80% of predicted.
  * FEV1/VC > 0.7.
  * Absence of active infection in the respiratory tract, documented with investigations directed by clinical symptoms, such as chest radiographs or computed tomographic scans or microbiologic cultures (sinus aspiration, upper respiratory tract viral screen, sputum culture, bronchoalveolar lavage) or active non-infectious lung disease (such as interstitial lung disease) that explain spirometric changes or chest CT findings.

Inclusion Criteria for Cohort B:

-Diagnosis of BOS-0p

* Decline in FEV1 of 10% - 19% of predicted compared with pretransplant testing OR
* Decline in predicted FEF25-75% (Forced Expiratory Flow between 25% and 75% of vital capacity) > 25%

Inclusion Criteria for Cohorts A and B:

* Age ≥18 years. Belumosudil is currently being tested in pediatric populations and the safety and efficacy in pediatric patients have not yet been established. A protocol amendment to include pediatric patients will be considered once safety in pediatric patients is established.
* ECOG performance status ≤2 (Karnofsky ≥ 60%).
* Participants must have adequate organ and marrow function as defined below:

  * WBC ≥ 3,000/μL
  * Absolute neutrophil count ≥ 1,500/ μL
  * Platelets ≥ 50,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤ 5 × institutional ULN
* No evidence of relapsed malignancy at the time of enrollment. Formal re-staging is not required for trial entry.
* All females of childbearing potential must have a negative serum or urine pregnancy test < 7 days before study drug administration.
* The ability to understand and willingness to sign a written consent document.

Exclusion Criteria for Cohorts A and B:

* Participants who have received prior therapy specifically for BOS. Therapy for cGVHD in the absence of BOS is permissible.
* Prior exposure to belumosudil.
* Participants who are receiving any other investigational immunosuppressive agents for cGVHD.
* Presence of an active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persistent fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Known human immunodeficiency virus infection. Interactions between belumosudil and anti-retroviral agents have not been established.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive. Subjects with previous positive serology results must have negative polymerase chain reaction results. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
24-week Overall Response Rate (ORR) [Cohort A] | up to 24 weeks.
  24-week ORR defined as the proportion of participants achieving BOS complete response (CR) or partial response (PR) based on change in FEV1 measurement per criteria of the 2014 NIH Consensus Conference.
24-week Overall Response Rate (ORR) [Cohort B] | up to 24 weeks.
  24-week ORR defined as the proportion of participants achieving BOS complete response (CR) or partial response (PR) based on change in FEV1 measurement per criteria of the 2014 NIH Consensus Conference.
24-week Progression Rate [Cohort B] | up to 24 weeks.
  24-week progression rate is defined as the proportion of participants experiencing BOS progression based on change in FEV1 measurement per criteria of the 2014 NIH Consensus Conference.

SECONDARY OUTCOMES:
48-weeks Overall Response Rate (ORR) [Cohort A] | Evaluated every 8 weeks, up to 48 weeks.
  48-week ORR defined as the proportion of participants achieving BOS complete response (CR) or partial response (PR) based on change in FEV1 measurement per criteria of the 2014 NIH Consensus Conference.
48-week Progression Rate [Cohort B] | Evaluated every 8 weeks, up to 48 weeks.
  48-week progression rate is defined as the proportion of participants experiencing BOS progression based on change in FEV1 measurement per criteria of the 2014 NIH Consensus Conference.
Grade 3-5 Treatment-Related Toxicity Rate | Evaluated on cycle 1 day 15, cycle 2, 3, 5, 7, 9, 11 (cycle duration=4 weeks) and end of treatment. Observed on treatment up to 12 cycles (48 weeks).
  All grade 3-5 AEs with attribution of probably, possibly or definitely-related to treatment based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Chronic Graft Versus Host Disease (cGVHD) Response | Evaluated every 8 weeks, up to 48 weeks.
  cGVHD response will be evaluated using non-pulmonary measurements per criteria of the 2014 NIH Consensus Conference.
Lee Symptom Scale (LSS) Quality of Life (QOL) Score | Evaluated on cycle 1 day 15, cycle 2, 3, 5, 7, 9, 11 (cycle duration=4 weeks) and end of treatment. Observed on treatment up to 12 cycles (48 weeks).
  Mean and standard deviation Lee Symptom Scale Quality of Life score estimated at each assessment timepoint. The LSS QOL scale is a 30-item measure with answers ranging from 0 "Not at All" to 4 "Extremely." Higher scores indicate greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu